CLINICAL TRIAL: NCT00313833
Title: A Randomized, Double Blind, Pilot Evaluation of the Effectiveness of BTDS Versus Placebo on Health Outcomes Associated With Analgesic Management of Elderly Residents in Supervised Living Environments
Brief Title: Safety and Effectiveness of Buprenorphine Transdermal System in Elderly Subjects With Chronic Pain: Pilot Study.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3002
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-04

CONDITIONS: Chronic Pain
Keywords: Chronic pain; elderly; supervised living; opioid; transdermal
MeSH Terms: conditions — Chronic Pain

INTERVENTIONS:
Drug: Buprenorphine transdermal delivery system

SUMMARY:
This pilot study was designed to evaluate the effectiveness and tolerability of the buprenorphine transdermal system versus placebo on health outcomes in elderly residents in supervised living environments. The treatment intervention duration is 42 days during which time supplemental analgesic medication (usual analgesic care) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain. Transdermal systems may offer advantages over currently indicated oral products including ease and convenience of use, improved compliance, possible reduction in patient care, and prolonged and consistent delivery of drug.

ELIGIBILITY:
Inclusion Criteria:

* residing in a nursing home, assisted living environment, or any type of supervised living situation in which the principal investigator maintained primary responsibility for the analgesic management of the resident.
* chronic pain of musculoskeletal origin who had been managed with short-acting opioids.

Exclusion Criteria:

* taking >90 mg oral morphine sulfate per day (during any single day) or >50 mcg/hr of transdermal fentanyl or its equivalent.
* activity restricted totally to bed rest.
* have cancer-related pain.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-12; Study Completion 2001-11

PRIMARY OUTCOMES:
Pilot study.

SECONDARY OUTCOMES:
The following outcome variables were assessed:
average pain intensity in the last 24 hours
acceptability of analgesic therapy
number of nighttime awakenings due to pain last night
quality of sleep
bowel status during the last 24 hours
pain management evaluation
symptom evaluation
staff evaluation of functional independence
resident-defined activity impairment scale
treatment satisfaction questionnaire
Health Assessment Questionnaire
Timed "Up & Go" evaluation
trail making test
digit span test
end of study global evaluation of therapeutic response
modified mini-mental state
examination and geriatric depression scale.
The following measures of health resource utilization were assessed:
use of analgesic medications (usual care plus BTDS) by product type
use of analgesic medications (usual care plus BTDS) by medication and dosage form
use of pain-related adjuvant medications by product type
number of phone calls to physicians for pain management
number of physician visits for pain management
and use of medications for the treatment of drug-related adverse events.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Birmingham Health Center, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Associated Physicians of Southbury, Southbury, Connecticut
  - Life Care Home Health Services, Delray Beach, Florida
  - Ward Parkway Health Services, Leawood, Kansas
  - Atlantic Medical Group LLC, Baltimore, Maryland
  - Bortz Health Care of Warren, Warren, Michigan
  - Bio-Test Clinic, Springfield, Missouri
  - Glengariff Health Care Center, Glen Cove, New York
  - Kings Harbor Multicare Center, The Bronx, New York
  - Regency Manor, Columbus, Ohio
  - Associated Medical Services Inc, Oklahoma City, Oklahoma
  - Town Center Village, Portland, Oregon
  - Center for Pain Management, Altoona, Pennsylvania
  - LAS/Health and Wellness Center, Zelienople, Pennsylvania
  - Geriatric Associates of America Inc PA, Baytown, Texas
  - Wisconsin Veterans Home, King, Wisconsin